CLINICAL TRIAL: NCT01022996
Title: An Open-label, Single-arm Phase II Study of RAD001 in Patients With Relapsed/Refractory Classical Hodgkin Lymphoma
Brief Title: Study of RAD001 in Patients With Relapsed/Refractory Hodgkin Lymphoma That Has Progressed After High-dose Chemotherapy and Autologous Stem Cell Transplant and/or After Gemcitabine- or Vinorelbine- or Vinblastine-based Treatment.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001NUS65
Record Dates: First submitted 2009-11-25; First posted 2009-12-01 (Estimated); Results first posted 2016-04-06 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-04

CONDITIONS: Hodgkin Lymphoma
Keywords: Hodgkin's Lymphoma; Hodgkin Lymphoma; Hodgkin's Disease; Hodgkin Disease; Lymphoma; Lymphoproliferative Disorders; Neoplasms by Histological type; Lymphatic Diseases; Hemic and Lymphatic Diseases; Recurrent Lymphoma; Refractory Lymphoma; Relapsed Lymphoma; Classical Hodgkin Lymphoma; Classical Hodgkin's Disease; Nodular sclerosing Hodgkin Lymphoma; Mixed-cellularity Hodgkin Lymphoma; Lymphocyte-rich Hodgkin Lymphoma; Lymphocyte depleted Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease; Lymphoma; Lymphoproliferative Disorders; Neoplasms by Histologic Type; Lymphatic Diseases; Hemic and Lymphatic Diseases | interventions — Everolimus

ARMS (1):
- RAD001 (Experimental): Patients with a history of classical Hodgkin lymphoma (ie, nodular sclerosing, mixed cellularity, lymphocyte-rich, lymphocyte-depleted) whose disease had progressed after receiving high-dose chemotherapy with AHSCT (if eligible) and/or after therapy with a gemcitabine- or vinorelbine- or vinblastine-containing regimen, were enrolled into this study. All patients were assigned to a daily dose of everolimus 10 mg (two 5-mg tablets), selfadministered orally and continuously from Cycle 1 Day 1 (Visit 2) until progression of disease, unacceptable toxicity, death, or discontinuation from the study for any other reason.
  A treatment cycle consisted of 28 days.
  Interventions: Drug: Everolimus (RAD001)

INTERVENTIONS:
Drug: Everolimus (RAD001) — Everolimus (RAD001) 10 mg (two 5mg tablets) given orally once daily and packed in blisters.
  Other Names: RAD001

SUMMARY:
This study will assess RAD001 in patients with refractory or relapsed Hodgkin Lymphoma that has progressed after high-dose chemotherapy and Autologous Stem cell transplant and/or after gemcitabine- or vinorelbine- or vinblastine-based treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of classical Hodgkin's lymphoma that has progressed after high-dose chemotherapy and Autologous Stem cell transplant and/or after gemcitabine- or vinorelbine- or vinblastine-based treatment
* Patients with at least one site of measurable disease measuring ≥ 2.0cm confirmed by PET and CT Scan (or MRI)
* Patients with adequate bone marrow, liver and renal function (confirmed by laboratory values)
* Patients with fasting serum cholesterol ≤300 mg/dL OR ≤7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN

Exclusion Criteria:

* Previous treatment with mTOR inhibitors
* Prior allogeneic stem cell transplant
* Chemotherapy, monoclonal antibody therapy, major surgery or treatment with other investigational drugs within 4 weeks of starting study treatment
* Another malignancy within 3 years of study entry (except adequately treated non-melanoma skin cancer and carcinoma in situ of the cervix)
* Severe and/or uncontrolled medical conditions that could affect participation in this study
* Female patients who are pregnant or breastfeeding; patients who are not willing to use adequate birth control during the study and for 8 weeks after the last study treatment Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2009-12; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (16):
- United States (16):
  - University of California at Los Angeles UCLS School of Medicine, Los Angeles, California
  - Rocky Mountain Cancer Centers RMCC - Aurora, Greenwood Village, Colorado
  - MD Anderson Cancer Center - Orlando, Orlando, Florida
  - Emory University School of Medicine/Winship Cancer Institute Emory University Med School, Atlanta, Georgia
  - Lurie Children's Hospital of Chicago Robert H. Lurie Comp Cancer, Chicago, Illinois
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute Karmanos-1, Detroit, Michigan
  - Mayo Clinic - Rochester Mayo Lymphoma Group, Rochester, Minnesota
  - Washington University School Of Medicine-Siteman Cancer Ctr StudyCoordinator:CLBH589B2201, St Louis, Missouri
  - New York Presbyterian Hospital Weill Cornell Med Ctr, New York, New York
  - Duke University Medical Center Duke University Medical Ctr, Durham, North Carolina
  - University of Tennessee Cancer Institute Univ Tennessee Cancer, Memphis, Tennessee
  - University of Texas/MD Anderson Cancer Center Dept.ofMDAndersonCancerCtr(3), Houston, Texas
  - University of Wisconsin Comprehensive Cancer Center Clinical Science Center - H4, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Johnston PB, Pinter-Brown LC, Warsi G, White K, Ramchandren R. Phase 2 study of everolimus for relapsed or refractory classical Hodgkin lymphoma. Exp Hematol Oncol. 2018 May 11;7:12. doi: 10.1186/s40164-018-0103-z. eCollection 2018. PMID 29774169
- See also: Related Info — http://NovartisClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- RAD001: Patients with a history of classical Hodgkin lymphoma (ie, nodular sclerosing, mixed cellularity, lymphocyte-rich, lymphocyte-depleted) whose disease had progressed after receiving high-dose chemotherapy with AHSCT (if eligible) and/or after therapy with a gemcitabine- or vinorelbine- or vinblastine-containing regimen, were enrolled into this study. Patients had at least one site of measurable disease at baseline ≥ 2.0 cm in the longest transverse diameter and clearly measurable in at least two perpendicular dimensions, as determined by CT scan. Patients received 10 mg of everolimus (two 5 mg tablets), self-administered orally once daily (qd), continuously from Cycle 1 Day 1 until progression of disease, unacceptable toxicity, death or discontinuation from the study for any other reason. The treatment cycle consisted of 28 days.
Period: Overall Study
Arm/Group | RAD001
Started | 57
Completed | 0
Not Completed | 57
Not completed — Adverse Event | 14
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 1
Not completed — Administrative problems | 6
Not completed — Disease Progression | 32
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) consisted of all patients who received at least 1 dose of study drug.
Arm/Group | RAD001
Number analyzed (Participants) | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.33 (14.101)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 24

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) Based on the Assessments by Investigator
Description: ORR: % of patients whose overall disease response was a complete response (CR) or a partial response (PR) in 8 cycles CR: Complete normalization of all index nodal & extranodal lesions: Radiological regression to normal size of all lymph nodes & nodal masses & complete disappearance of all lesions PR: At least a 50% decrease in the SPD of all index nodal & extranodal lesions FDG-avid or PET positive prior to therapy: one or more PET positive at previously involved site.At least a 50% increase in the SPD of all index nodal & extranodal lesions, taking as reference the smallest sum of the product of the diameters of all index lesions recorded at or after baseline . Lesions PET positive if FDG-avid lymphoma or PET positive prior to therapy. Unknown (UNK): Progression not documented & one or more of the index lesions not assessed or assessed using a different method than baseline at the time of radiologic evaluation. Each cycle was 28 days.
Time Frame: at screening and every threee months beginning at cycle 3 until end of treatment due to progression of disease, unacceptable toxicity, death or discontinuation from the study for any other reason
Population: Full analysis set (FAS) consisted of all patients who received at least 1 dose of study drug and was the primary set for efficacy analyses.
Measure: Number; unit: percentage of participants
Arm/Group | RAD001
Number analyzed (Participants) | 57
percentage of participants
  Complete response (CR) | 8.8
  Partial response (PR) | 36.8
  Response of CR or PR | 45.6

2. Secondary Outcome: Time to Overall Response (TTR) Per Kaplan-Meier Estimate
Description: Time to overall response was defined as the time from the first date of treatment to the date of first documented response of CR or PR. Time to overall response is applied to patients whose best overall response is CR or PR. Patients who drop-out or did not have a response (CR or PR) will be treated as censored at the date of last adequate tumor assessment.
Time Frame: Every three months beginning at Cycle 3 until end of treatment due to progression of disease, unacceptable toxicity, death or discontinuation from the study for any other reason
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | RAD001
Number analyzed (Participants) | 57
Days | NA [79.00 to NA] — N/A = Not achieved

3. Secondary Outcome: Duration of Overall Response (DoR)
Description: The duration of overall response was calculated from the date of first documented response (CR or PR) to the date of first documented disease progression or death due to any cause or start of a new antineoplastic therapy. This only applies to patients whose best overall response is CR or PR.
Time Frame: as for outcome 2
Population: Full analysis set (FAS): consisted of all patients who received at least 1 dose of study drug and was the primary set for efficacy analyses.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | RAD001
Number analyzed (Participants) | 57
Days | 350.8 (388.63)

4. Secondary Outcome: Disease Control Rate (DCR)
Description: The disease control rate was defined as the percentage of patients with a best overall response of CR, PR or stable disease (SD).
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RAD001
Number analyzed (Participants) | 57
Percentage of participants | 80.7 [68.09 to 89.95]

5. Secondary Outcome: Duration of Disease Control
Description: The duration of overall response (CR/PR) was applied only to patients whose best overall response was CR or PR. Duration of overall response was calculated from the date of the first documented response of CR or PR to the date of first documented disease progression or death due to any cause or start of a new antineoplastic therapy.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | RAD001
Number analyzed (Participants) | 57
Days | 321.9 (394.92)

6. Secondary Outcome: Progression Free Survival (PFS) by Kaplan-Meier Estimate
Description: Progression-free survival (PFS) was defined as the time from the first date of treatment to the date of first documented disease progression or death due to any cause or start of a new antineoplastic therapy. An event for PFS was defined as a documented disease progression or death due to any cause or start of a new antineoplastic therapy, whichever occurred first. Cycle = 28 days.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | RAD001
Number analyzed (Participants) | 57
Days | 8.0 [5.07 to 10.96]

ADVERSE EVENTS:
Arm/Group | RAD001
Serious Adverse Events (participants affected / at risk) | 18/57
Other Adverse Events (participants affected / at risk) | 56/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RAD001 (N=57)
Anaemia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Myocarditis (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Drug ineffective (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 3
Influenza (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 4
Pseudomembranous colitis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Haemoglobin decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Complex regional pain syndrome (Nervous system disorders) | 1
Nerve compression (Nervous system disorders) | 1
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 2
Subclavian artery occlusion (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RAD001 (N=57)
Anaemia (Blood and lymphatic system disorders) | 18
Neutropenia (Blood and lymphatic system disorders) | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 27
Vision blurred (Eye disorders) | 4
Abdominal distension (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 9
Abdominal pain upper (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 15
Dyspepsia (Gastrointestinal disorders) | 5
Mouth ulceration (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 14
Stomatitis (Gastrointestinal disorders) | 14
Toothache (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 13
Chest discomfort (General disorders) | 4
Chest pain (General disorders) | 6
Chills (General disorders) | 5
Fatigue (General disorders) | 33
Localised oedema (General disorders) | 3
Malaise (General disorders) | 3
Mucosal inflammation (General disorders) | 5
Oedema peripheral (General disorders) | 12
Pain (General disorders) | 7
Peripheral swelling (General disorders) | 3
Pyrexia (General disorders) | 18
Bronchitis (Infections and infestations) | 7
Nasopharyngitis (Infections and infestations) | 5
Oral herpes (Infections and infestations) | 3
Pneumonia (Infections and infestations) | 4
Rhinitis (Infections and infestations) | 4
Sinusitis (Infections and infestations) | 10
Upper respiratory tract infection (Infections and infestations) | 14
Urinary tract infection (Infections and infestations) | 4
Contusion (Injury, poisoning and procedural complications) | 4
Alanine aminotransferase increased (Investigations) | 8
Aspartate aminotransferase increased (Investigations) | 9
Blood alkaline phosphatase increased (Investigations) | 9
Blood cholesterol increased (Investigations) | 3
Blood glucose increased (Investigations) | 3
Blood lactate dehydrogenase increased (Investigations) | 6
Liver function test abnormal (Investigations) | 3
Weight decreased (Investigations) | 7
White blood cell count decreased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 7
Hypercholesterolaemia (Metabolism and nutrition disorders) | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 10
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 7
Hypocalcaemia (Metabolism and nutrition disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Back pain (Musculoskeletal and connective tissue disorders) | 15
Joint swelling (Musculoskeletal and connective tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8
Dysgeusia (Nervous system disorders) | 8
Headache (Nervous system disorders) | 13
Neuropathy peripheral (Nervous system disorders) | 9
Anxiety (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 27
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3
Acne (Skin and subcutaneous tissue disorders) | 8
Night sweats (Skin and subcutaneous tissue disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 12
Rash (Skin and subcutaneous tissue disorders) | 22
Hot flush (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.